CLINICAL TRIAL: NCT01701518
Title: A Prospective Multicentre Pilot Study of the Effectiveness of an Intra-operative Intravitreal Sustained Release Dexamethasone Implant (Ozurdex®) in Vitrectomy Surgery for Epiretinal Membranes
Brief Title: A Pilot Study of the Effectiveness of Intra-operative Ozurdex® in Vitrectomy Surgery for Epiretinal Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other); Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZ123; OZ123 (Other: Health Canada)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Epiretinal Membrane; Macular Edema
Keywords: Ozurdex; Dexamethasone; Epiretinal membrane; Macular edema
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ozurdex (Other): Intra-operative Ozurdex (biodegradable 0.7mg dexamethasone implant) post-vitrectomy for epiretinal membrane
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Ozurdex — biodegradable 0.7mg dexamethasone implant
  Other Names: 0.7mg dexamethasone implant

SUMMARY:
To determine if an intravitreal sustained release dexamethasone implant (Ozurdex®) injected at the conclusion of surgery in patients undergoing vitrectomy and membrane peeling for idiopathic epiretinal membranes is safe and effective to decrease the macular edema, as demonstrated by a gain in vision and decreased in retinal thickness and volume.

DETAILED DESCRIPTION:
We believe that the use of intravitreal corticosteroids post-operatively has the capacity to mitigate much of the residual swelling and retinal thickening that is seen after vitrectomy for epiretinal membranes. The unique pharmacokinetics of the sustained released dexamethasone implant (Ozurdex®) makes it an ideal delivery system to use post-vitrectomy for epiretinal membrane surgery. Its duration of action and its drug delivery characteristics over 6 months approximately match the post-operative time course of healing and remodeling in an edematous retina.

This is a prospective, multicentre, pilot study evaluating the efficacy of an intravitreal sustained release dexamethasone implant (Ozurdex®) injected at the conclusion of surgery in 15 patients undergoing vitrectomy and membrane peeling for idiopathic epiretinal membranes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vitrectomy surgery for a visually significant (≤ 20/50) idiopathic epiretinal membrane.
* Central retinal thickness ≥ 250 μm.
* Age more than 18 years old.
* Decision makers able to give informed consent.
* Females of child bearing potential must agree to use acceptable means of birth control for the duration of the study.

Exclusion Criteria:

* Secondary epiretinal membranes (ex: secondary to a retinal vein occlusion, etc.).
* Any other macular pathology that could affect anatomic or functional results.
* History of uveitis requiring intravitreal triamcinolone injection.
* History of steroid-responsive glaucoma.
* History of moderate or advanced glaucoma (cup to disc ratio ≥ 0.7).
* IOP > 23 mm Hg if untreated, or > 21 mm Hg if treated with medication.
* Pregnant or breast-feeding woman.
* Unable to attend the scheduled follow-up appointments.
* Patients with known hypersensitivity to any components of Ozurdex® or to other corticosteroids.
* Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 3 Months
  Best corrected visual acuity measured before surgery and 3 months after surgery using an early treatment diabetic retinopathy study (ETDRS) chart.

SECONDARY OUTCOMES:
Best corrected visual acuity at 1,4 and 6 months | 6 months
  Best corrected visual acuity measured at 1,4 and 6 months after surgery using an early treatment diabetic retinopathy study (ETDRS) chart.
Retinal thickness and volume | 6 months
  Measure the change in retinal thickness and volume from baseline and at 1, 3, 4, 6 months using optical coherence tomography (OCT).
Intraocular pressure (IOP) | 6 months
  Change of IOP from baseline will be monitored.
Cataract progression (if applicable) | 6 months
  For phakic patients, cataract progression from baseline to the 6 months visit will also be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Kertes, MD,CM,FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario